CLINICAL TRIAL: NCT00976690
Title: A Multicentre Randomized Open Study Comparing Azathioprine to Mesalazine for the Prevention of Postoperative Recurrence in the Crohn Disease
Brief Title: Comparison Azathioprine to Mesalazine for the Prevention of Postoperative Recurrence in the Crohn Disease
Acronym: IMURELPOST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2001-1
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Crohn Disease
Keywords: Crohn's Disease; Ileocolic resection; Endoscopic recurrence; Ileocolic or colon resection (>50cm)
MeSH Terms: conditions — Crohn Disease | interventions — Azathioprine; Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Azathioprine : 2mg/kg/day
  Interventions: Drug: Azathioprine OR Mesalazine
- 2 (Active Comparator): Mesalazine : 4g/day
  Interventions: Drug: Azathioprine OR Mesalazine

INTERVENTIONS:
Drug: Azathioprine OR Mesalazine — Azathioprine : 2mg/kg/day Mesalazine : 4g/day

SUMMARY:
To show the superiority of Azathioprine comparing Mesalazine in the prevention of postoperative recurrence in Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* Clinical remission at inclusion time (CDAI<150)
* Having ileocolonic or colon resection 21 days before inclusion
* Resection > 50cm or subtotal colectomy with ileorectal anastomosis

Exclusion Criteria:

* Intolerance to one of both study treatment
* Liver failure (TP<60%)
* Renal Failure (Creatinine < Lab results)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2002-10; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinically and endoscopically recurrence at 12 and 24 months | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc LEMANN, MD,PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (14):
- France (14):
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - CHU CAEN, Caen
  - Hopital Beaujon, Clichy
  - Chru Lille, Lille
  - Hopital Lariboisiere, Paris
  - Hopital Saint Louis, Paris
  - Hopital St Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Haut Leveque, Pessac
  - Chu Reims, Reims
  - Chu Rennes, Rennes
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours

REFERENCES:
- See also: Related Info — http://www.getaid.org